CLINICAL TRIAL: NCT04538495
Title: Characterization of Multisystem Inflammatory Syndrome in Children (MIS-C) and Its Relationship to Kawasaki Disease
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jane C. Burns MD, Principal Investigator, University of California, San Diego
Other Study IDs: CER-1602-34473
Record Dates: First submitted 2020-08-19; First posted 2020-09-04 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2021-11

CONDITIONS: Kawasaki Disease; Inflammation
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome; Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 12.5 cc of blood (2.5 teaspoons) (for RNA studies, plasma protein studies, serum antibody measurement, and in vitro studies of PBMC and cultured HUVECs) will be drawn when phlebotomy is performed for routine clinical care from MIS-C. This will be at 3 timepoints: admission (pre-treatment), after treatment but before discharge, at the clinic visit between 1 to 6 weeks after discharge. Whole blood RNA will be collected in PAXgene tubes.
  Rectal swab or stool for SARS-CoV-2 PCR testing in the Burns Lab at UCSD will be collected only once at the time of admission.
  For sites able/willing to participate in live cell collection, heparinized blood (green top tubes) for PBMC and neutrophil studies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Beginning in mid-March 2020, pediatricians in communities in Western Europe, the UK, and the Eastern U.S. that had been severely affected by the Covid-19 pandemic noted an increased number of children presenting with fever and evidence of severe inflammation who required admission to intensive care. The syndrome was branded by the CDC in the U.S. as Multisystem Inflammatory Syndrome in Children (MIS-C). The most severely affected children presented with heart failure leading to shock and the absence of significant pulmonary disease. The clinical presentation in these patients shared many features with Kawasaki disease (KD), a self-limited pediatric vasculitis that can result in coronary artery aneurysms.The inflammatory markers, however, were much higher even than KD shock syndrome, a variant of KD presenting with distributive shock and requiring inotropic and vasoactive support in the ICU. Some patients were polymerase chain reaction (PCR)+ for SARS-CoV-2 while most were virus-negative but had detectable antibody suggesting that MIS-C was an immune-mediated reaction to antecedent exposure to the virus. While patients were being diagnosed with shock and MIS-C, children with a milder version of MIS-C that shared many features of KD were being diagnosed in these same regions.

DETAILED DESCRIPTION:
Clinical characterization (Burns, Tremoulet, Sivilay, Roberts, Jain): Over the 8 months of enrollment funded by this supplement, 30 sites will collect data on KD and MIS-C patients using the detailed case report form in our REDCap database. This includes data on patient demographics, clinical presentation, laboratory data, treatments, clinical outcomes, and cardiovascular outcomes on all KD and MIS-C patients so that the investigators can develop a systematic picture of the different patient groups (see details below).

Parent observations (Kim): To learn about signs and symptoms in the patient and family members leading up to acute presentation a parent questionnaire will be devised and analyzed by Dr. Katherine Kim with the Patient and Parent Advisory Board. The investigators will collect known signs and symptoms as well as those that may not have been previously reported in the literature and record presence/absence, location in the body, and severity level by day. The questionnaire will be available as a mobile/web application and via paper. With these data, the investigators will conduct an exploratory analysis to characterize symptom phenotypes and the relationships of these profiles with demographic features and clinical characteristics. In addition, the investigators will assess whether we can detect differences between the symptom phenotypes of KD and MIS-C. The investigators will conduct cluster analysis to identify symptom phenotypes from aggregate symptom observations blinded as to presumed or verified diagnosis (n=100 with each sign/symptom on each day as a distinct data point). Phenotypes may include characteristics such as symptoms that co-occur or are independent, and symptom burden index (e.g., number symptoms present). The investigators will use Ward's hierarchical cluster analysis to estimate the number of likely clusters.3 The investigators will apply K-means nonhierarchical cluster analysis repeated 100 times in a leave-one out validation model to assure repeatability and stability within the model. The investigators will create score indices analyzed with logistic regression, principal component analysis, factor analysis and correlation analysis. The investigators will then assess whether clusters are related to verified diagnosis and/or sociodemographic characteristics such as age, race/ethnicity, geography. The investigators will use discriminant analysis techniques and more recent classification techniques such as CART to examine if symptom phenotypes of KD and MIS-C are dissimilar. If information in terms of symptom clusters at a point in time or a trajectory of a single symptom over time are insufficient to distinguish between the two conditions, this would provide support for the argument that the recorded symptoms are insufficient for discrimination or that the two disease entities are not symptomatically different. This exploratory analysis will provide important information that can be further developed for clinical guidance and parent education.

Photography (Kim, Tremoulet): Patient photographs of the eye, mouth/tongue, and rash will be collected as a novel addition to the usual clinical data. These photographs obtained before treatment will document the presence or absence of conjunctival injection and perilimbal sparing, mucocutaneous changes in the oropharynx including changes in the vermillion border (erythema, fissuring) and the tongue (strawberry tongue), and the nature of the rash. The photographs will be subjected to analysis using facial recognition software and artificial intelligence approaches used by our collaborators at the University of Southern California Center for Artificial Intelligence in Society led by Hayden Shively and Lucas Hu to evaluate whether a computer algorithm can be created that can differentiate the clinical characteristics of MIS-C from photographs taken of children with acute KD and those with other pediatric febrile illnesses. Dr. Katherine Kim at UC Davis will compare the photos with the questionnaire responses to supplement the parent descriptions of signs and symptoms and validate the observations. This comparison can result in enhanced descriptions using the words of parents themselves. Photography is needed to document these physical findings as the investigators have learned over the years that physician description of these features is woefully inaccurate. The finding, for example, of a strawberry tongue is a specific injury pattern that involves sloughing of the cornified tips of the filiform papillae and has historically been associated with only 3 conditions: staphylococcal and streptococcal toxin-mediated disease and KD.

ELIGIBILITY:
Inclusion criteria:

The following patients (age 1 mos. through young adults) will be recruited for this study:

Patients who meet the CDC definition for MIS-C:

* Patients presenting with fever (>38C for >24 h - also by subjective report), laboratory evidence of inflammation, and evidence of clinically severe illness requiring hospitalization, with multisystem (>2) organ involvement (cardiac, renal, respiratory, hematologic, gastrointestinal, dermatologic or neurological); AND
* No alternative plausible diagnoses; AND Positive for current or recent SARS-CoV-2 infection by RT-PCR, serology, or antigen test; or suspected COVID-19 exposure within the 4 weeks prior to the onset of symptoms
* Patients who meet the CDC definition for MIS-C and require care in the PICU

Exclusion Criteria:

• All patients with pre-existing major medical conditions will be excluded. This includes patients with known genetic disorders (e.g. trisomy 21, cystic fibrosis), conditions requiring continuous medication (e.g. seizure disorder, heart disease), or known immune disorder (e.g. hypogammaglobulinemia, complement deficiency). Patients with asthma or atopic dermatitis will not be excluded unless patients have received oral steroids in the previous week. Obesity is not an exclusion.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We plan to enroll 100 MIS-C subjects in this study to allow for the collection of data and samples that will support the many different aims in this study.
Sampling Method: Non-Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Collection of clinical data and patient samples from children with MIS-C and KD to | We will collect demographic and clinical data on all KD patients at participating sites throughout the 8-month study period.
  Collection of clinical data and patient samples from children with MIS-C and KD to understand the relationship between these two conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Jane C Burns, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No